CLINICAL TRIAL: NCT05477511
Title: The Effect of in Utero Hyperglycaemia, Maternal Overnutrition and Interaction With Postnatal Lifestyle on Cardiometabolic Risk at Young Adulthood - Extension of HAPO Follow-up Study
Brief Title: The Extension of HAPO Follow-up Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ronald Wang, Professor, Chinese University of Hong Kong
Other Study IDs: HAPO-005
Record Dates: First submitted 2022-07-21; First posted 2022-07-28 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Hyperglycemia; Pregnancy; Overnutrition; Maternal Obesity During Childbirth; Diabetes Mellitus; Cardiovascular Diseases; Gestational Diabetes Mellitus in Pregnancy; Hypertension
Keywords: Hyperglycemia; Pregnancy; Overnutrition; Maternal Obesity; Diabetes Mellitus; Cardiovascular Diseases; Gestational Diabetes Mellitus; Hypertension; Young Adulthood
MeSH Terms: conditions — Hyperglycemia; Overnutrition; Diabetes Mellitus; Cardiovascular Diseases; Hypertension; Pregnancy in Obesity; Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Fasting blood, OGTT blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mother: Chinese mother in Hong Kong who had been assessed in HAPO follow-up study when their children was at either 7 or 11-14 years of age
- 18 years old child of the enrolled mother: Children who had been assessed in HAPO follow-up study at either 7 or 11-14 years of age

SUMMARY:
The prevalence of diabetes mellitus (DM) and cardiovascular disease (CVD) escalate remarkably worldwide and obesity becomes an epidemic disease. This study is interested in how the model of Developmental Origin of Health and Disease (DOHaD) influence individual's health status as they reach young adulthood. Since the mothers from HAPO study have not been subjected to antenatal treatment on the various degree of maternal hyperglycaemia in pregnancy, this would be an unique cohort that allows determination of the effect of various degree of maternal hyperglycaemia below the level of overt DM, on children's cardiometabolic risk in Chinese population.

DETAILED DESCRIPTION:
The investigators recruited 1760 Chinese pregnant women between 2000 and 2005. The HAPO study investigated whether any adverse outcome was associated with mild degree of GDM. All mothers underwent a 75-gram OGTT at 24-32 weeks gestation, but clinicians were blinded to the results as long as the fasting PG was ≤ 5.8 mmol/L & 2-hour PG ≤ 11.1 mmol/L. The maternal serum C-peptide and HbA1c, cord serum C-peptide and early neonatal PG, pregnancy outcome and the neonatal anthropometric parameters are available for future study. This is so far the largest cohort in a Chinese population who has been investigated for glycaemia during pregnancy, but with OGTT results remained undisclosed to subjects and clinicians. This unique cohort can allow us to study the effect of in-utero hyperglycemia on the cardiometabolic risks at childhood, adolescence and adulthood.

Eligible subjects are all mother-child pairs participating in the original HAPO study. Children born preterm before 37 weeks of gestation, non-Chinese and whose mother's OGTT result were unblinded during pregnancy will be excluded.The family (the child and the mother) will be invited for a third follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Mother-child pairs who had been assessed in HAPO follow-up study at either 7 years or 11-14 years old

Exclusion Criteria:

* Children born preterm before 37 weeks of gestation
* Non-Chinese
* Mothers' OGTT results were unblinded during pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Hong Kong women and their 18 year-old offspring
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2020-08-28 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of DM in the young adult offspring | At a time around 18 years of age
  Study specimens would be collected to identify the rate of DM in young adult offspring.

SECONDARY OUTCOMES:
Rate of impaired glucose regulation, obesity and adiposity, hypertension and various insulin indices | At a time around 18 years of age
  Study specimens would be collected to identify the percentage of impaired glucose regulation, obesity and adiposity, hypertension and various insulin indices in young adult offspring.

CONTACTS AND LOCATIONS:
Overall Officials: Chi Chiu Wang, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong, China, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] See protocol

DOCUMENTS (1):
  • Study Protocol (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/11/NCT05477511/Prot_000.pdf